CLINICAL TRIAL: NCT03428100
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Safety and Efficacy of Baricitinib in Combination With Topical Corticosteroids in Adult Patients With Moderate-to-Severe Atopic Dermatitis Who Have Experienced Failure to Cyclosporine or Are Intolerant to, or Have Contraindication to, Cyclosporine
Brief Title: A Long-term Study of Baricitinib (LY3009104) With Topical Corticosteroids in Adults With Moderate to Severe Atopic Dermatitis That Are Not Controlled With Cyclosporine or for Those Who Cannot Take Oral Cyclosporine Because it is Not Medically Advisable
Acronym: BREEZE-AD4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16841; I4V-MC-JAIN (Other: Eli Lilly and Company); 2017-004574-34 (EudraCT Number)
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04-15

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (19):
- 4 mg Baricitinib (Experimental): 4 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- 2 mg Baricitinib (Experimental): 2 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- 1 mg Baricitinib (Experimental): 1 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- Placebo (Placebo Comparator): Placebo administered orally once daily in combination with topical corticosteroids. Additional Placebo administered orally to maintain the blind.
  Interventions: Drug: Placebo; Drug: Topical corticosteroid
- Long Term Extension(LTE) Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) (Experimental): 4 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) (Experimental): 4 mg Baricitinib rerandomized to 2 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) (Experimental): 2 mg Baricitinib rerandomized to 2 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders) (Experimental): 2 mg Baricitinib rerandomized to 1 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (Experimental): 4 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (Experimental): 2 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (Experimental): 1 mg administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy (Placebo Comparator): Placebo administered orally once daily (continued previous dose) in combination with topical corticosteroids. Additional placebo administered orally to maintain the blind.
  Interventions: Drug: Placebo; Drug: Topical corticosteroid
- LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): 4 mg administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): 2 mg Baricitinib rerandomized to 2 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): 2 mg Baricitinib rerandomized to 4 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): 1 mg Baricitinib rerandomized to 2 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): 1 mg Baricitinib rerandomized to 4 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): Placebo rerandomized to 2 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid
- LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (Experimental): Placebo rerandomized to 4 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo; Drug: Topical corticosteroid

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 1 mg Baricitinib; 2 mg Baricitinib; 4 mg Baricitinib; LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy; LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy; LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy; LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy; LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders); LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders); LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders); Long Term Extension(LTE) Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders)
Drug: Placebo — Administered orally.
Drug: Topical corticosteroid — Administered as standard-of-care.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of baricitinib in combination with topical corticosteroids in participants with moderate to severe atopic dermatitis who have experienced failure to cyclosporine or are intolerant to, or have contraindication to cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with moderate to severe Atopic Eczema (Atopic Dermatitis) for at least 12 months.
* Have had inadequate response to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.
* Have a medical contraindication to cyclosporine, or had intolerance and/or unacceptable toxicity or inadequate response to cyclosporine in the past.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episodes of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or are currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * Monoclonal antibody for less than 5 half-lives prior to randomization.
  * Received prior treatment with any oral Janus kinase (JAK) inhibitor less than 4 weeks prior to randomization.
  * Received oral corticosteroids within 4 weeks prior to randomization or parenteral corticosteroids administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study.
  * Have had an intra-articular corticosteroid injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization.
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of recurrent (≥ 2) VTE or are considered at high risk of VTE as deemed by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent and/or clinically serious viral, bacterial, fungal, or parasitic infection including but not limited to herpes zoster, tuberculosis.
* Have specific laboratory abnormalities related to thyroid, renal and liver function, or blood cells.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (103):
- Austria (5):
  - Universitätsklinikum Graz, Graz, Styria
  - Universitätsklinik Innsbruck, Innsbruck, Tyrol
  - KA Rudolfstiftung, Vienna
  - AKH, Vienna
  - Sozialmed. Zentrum Ost - Donauspital, Vienna
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven - Campus Sint-Rafaël, Leuven
- Brazil (9):
  - Cedoes Centro Diagnostico Pequisa Osteoporose E Santo Ltd, Vitória, Espírito Santo
  - CCBR Brasil Centro de Analises e Pesquisas Clínicas LTDA, Rio de Janeiro, Rio de Janeiro
  - IDERJ - Instituto de Dermatologia e Estética do Brasil, Rio de Janeiro, Rio de Janeiro
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento - Instituto de Educação e Pesquisa, Porto Alegre, Rio Grande do Sul
  - Faculdade de Ciências Médicas - UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas da FMRP, Ribeirão Preto, São Paulo
  - Fundação Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital da Clinicas da Faculdade de Medicina da USP, São Paulo
- Finland (3):
  - Terveystalo Tampere, Tampere, Irkanmaa
  - Helsinki University Central Hospital, Helsinki
  - Hospital Mehiläinen Neo, Turku
- France (10):
  - Hôpital de Pontchaillou, Rennes, Cedex 9
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - CHU de Bordeaux Hopital Saint Andre, Bordeaux
  - Hôpital C. HURIEZ, Lille
  - Hôpital Emile Muller, Mulhouse
  - Chru De Nantes Hotel-Dieu, Nantes
  - CHU de Nice Hopital de L'Archet, Nice
  - Hopital Sainte Anne (H.I.A), Toulon
  - Hopital Larrey, Toulouse
  - Centre Hospitalier de Valence, Valence
- Germany (17):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Hautarztpraxis Dr. Leitz und Kollegen, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Rechts der Isar der TU München, München, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Elbe Kliniken Stade Buxtehude GmbH Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Klinische Forschung Osnabrück, Osnabrück, Lower Saxony
  - Fachklinik Bad Bentheim, Bad Bentheim, North Rhine-Westphalia
  - St Josef-Hospital Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
- Italy (10):
  - Fondazione IRCCS Osp.Maggiore Policlinico - Dermatologia, Milan, Milan
  - Ospedale Clinicizzato San Donato, San Donato Milanese, Milan
  - Dip.to Med. Sperimentale -Polic.Umberto I -Univ. La Sapienza, Roma, Rome
  - Azienda Ospedaliera Umberto I, Ancona
  - Spedali Civili - Universita degli Studi, Brescia
  - Fondazione Universitaria degli Studi G D'Annunzio, Chieti
  - Azienda Ospedaliera di Perugia, Perugia
  - Arcispedale Santa Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Policlinico di Tor Vergata, Roma
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
- Japan (11):
  - Yanagihara dermatology clinic, Ainokawa, Ichikawa-shi, Chiba
  - Fumimori Clinic, Fukuoka, Fukuoka
  - Queen's Square Dermatology and Allergology, Nishi-ku, Yokohama-city, Kanagawa
  - Noguchi Dermatology, Kashima-machi, Kamimashiki-gun, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Kume Clinic, Nishi-ku Sakai-shi, Osaka
  - Sanrui Dermatology Clinic, Ohmiya-ku,Saitama-shi, Saitama
  - Iidabashi Clinic, Chiyoda-ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Bravis Ziekenhuis, Bergen op Zoom
  - Amphia Ziekenhuis, Breda
- Poland (10):
  - NZOZ Specjalistyczna Przychodnia Dermatologiczna Specderm, Bialystok
  - Centrum Badan Klinicznych, PI House, Gdansk
  - Centrum Medyczne Angelius Provita, Katowice
  - Barbara Rewerska DIAMOND CLINIC, Krakow
  - Dermed Centrum Medyczne Sp. z o.o., Lodz
  - Miejski Szpital Zespolony w Olsztynie Klinika Dermatologii, Olsztyn
  - DermoDent, Centrum Medyczne Czajkowscy, Osielsko
  - LASER CLINIC Specjalistyczne Gabinety Lekarskie, Szczecin
  - Centralny Szpital Kliniczny MSW Klinika Dermatologii, Warsaw
  - Wojskowy Instytut Medyczny CSK MON, Warsaw
- Russia (5):
  - State scientific centre for dermatovenerology and cosmetolog, Moscow
  - First Moscow State Medical University n.a. Sechenov, Moscow
  - SPb SBHI Skin-venerologic dispensary #10, Saint Petersburg
  - LLC ArsVitae NorthWest, Saint Petersburg
  - LLC Medical Center "Kurator", Saint Petersburg
- Spain (7):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Univ. Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Hospital de Manises, Manises, Valencia
  - Hospital De Basurto, Bilbao, Vizcaya
  - Hospital Universitario Dr Pesset, Valencia
- Switzerland (3):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Bern, Bern
  - Universitätsspital Zürich, Zurich
- United Kingdom (6):
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - West Glasgow Ambulatory Care Hospital, Glasgow, Lanarkshire
  - Whipps Cross University Hospital, Leytonstone, London
  - Broadgreen Hospital, Liverpool, Merseyside
  - Guys/St. Thomas Hospital, London, Surrey
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Katoh N, Takita Y, Isaka Y, Nishikawa A, Torisu-Itakura H, Saeki H. Pooled Safety Analysis of Baricitinib in Adult Participants with Atopic Dermatitis in the Japanese Subpopulation from Six Randomized Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2765-2779. doi: 10.1007/s13555-022-00828-5. Epub 2022 Oct 18. PMID 36255569
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- See also: A Long-term Study of Baricitinib (LY3009104) With Topical Corticosteroids in Adults With Moderate to Severe Atopic Dermatitis (Eczema) Not Controlled With Cyclosporine or for Those Who Cannot Take Oral Cyclosporine Because it is Not Medically Adv — https://www.lillytrialguide.com/en-US/studies/eczema/JAIN#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg Baricitinib: 1 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  .
- LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy: 1 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
- LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy: 4 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Period: Double-Blind Treatment Week 0 to Week 52
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Long Term Extension(LTE) Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders) | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy | LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy
Started | 93 | 93 | 185 | 92 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 93 | 93 | 184 | 92 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 72 | 80 | 173 | 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 21 | 13 | 12 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 16 | 10 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Extension Week 52 to Week 200
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Long Term Extension(LTE) Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders) | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy | LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy
Started | 0 (Participants who completed the study through Week 52 progressed to the Long-term Extension Phase.) | 0 (Participants who completed the study through Week 52 progressed to the Long-term Extension Phase.) | 0 (Participants who completed the study through Week 52 progressed to the Long-term Extension Phase.) | 0 (Participants who completed the study through Week 52 progressed to the Long-term Extension Phase.) | 16 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization, were receiving investigational product, and had not used high- or ultra-high-potency TCS in the previous 14 days were enrolled into the downtitration substudy.) | 16 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization, were receiving investigational product, and had not used high- or ultra-high-potency TCS in the previous 14 days were enrolled into the downtitration substudy.) | 25 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization, were receiving investigational product, and had not used high- or ultra-high-potency TCS in the previous 14 days were enrolled into the downtitration substudy.) | 24 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization, were receiving investigational product, and had not used high- or ultra-high-potency TCS in the previous 14 days were enrolled into the downtitration substudy.) | 7 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who received Baricitinib 4 mg, 2 mg, 1 mg or placebo and were not eligible for the randomized downtitration substudy remained on their current dose of Baricitinib. If worsening of the symptoms occurred (IGA is ≥3), those receiving Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 22 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who received Baricitinib 4 mg, 2 mg, 1 mg or placebo and were not eligible for the randomized downtitration substudy remained on their current dose of Baricitinib. If worsening of the symptoms occurred (IGA is ≥3), those receiving Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 34 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who received Baricitinib 4 mg, 2 mg, 1 mg or placebo and were not eligible for the randomized downtitration substudy remained on their current dose of Baricitinib. If worsening of the symptoms occurred (IGA is ≥3), those receiving Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 29 (At Week 52: Responders (IGA 0 or 1) and partial responders (IGA 2) who received Baricitinib 4 mg, 2 mg, 1 mg or placebo and were not eligible for the randomized downtitration substudy remained on their current dose of Baricitinib. If worsening of the symptoms occurred (IGA is ≥3), those receiving Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 24 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 27 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 26 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 13 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 14 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 11 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.) | 12 (At Week 52: Nonresponders (IGA ≥ 3) in the Placebo, Baricitinib 2 mg or 1 mg were rerandomized (1:1) to Baricitinib 4 mg or 2 mg.)
Completed | 0 | 0 | 0 | 0 | 2 | 6 | 5 | 6 | 3 | 5 | 5 | 10 | 1 | 6 | 4 | 4 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 14 | 10 | 20 | 18 | 4 | 17 | 29 | 19 | 23 | 21 | 22 | 9 | 13 | 10 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 4 | 0 | 4 | 4 | 0 | 9 | 9 | 6 | 3 | 4 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 10 | 4 | 8 | 8 | 3 | 7 | 11 | 11 | 8 | 6 | 12 | 5 | 3 | 1 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 2 | 0 | 6 | 13 | 5 | 2 | 5 | 1 | 0 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Total
Number analyzed (Participants) | 93 | 93 | 185 | 92 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (13.6) | 38.9 (14.0) | 37.3 (13.6) | 38.7 (13.3) | 38.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 35 | 52 | 35 | 166
  Male | 49 | 58 | 133 | 57 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 26 | 14 | 64
  Not Hispanic or Latino | 54 | 62 | 101 | 55 | 272
  Unknown or Not Reported | 28 | 18 | 58 | 23 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 16 | 19 | 36 | 18 | 89
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 3 | 11
  White | 74 | 70 | 145 | 71 | 360
  More than one race | 0 | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 3 | 2 | 4 | 10
  Netherlands | 3 | 0 | 9 | 4 | 16
  Belgium | 3 | 5 | 12 | 6 | 26
  Finland | 2 | 2 | 2 | 1 | 7
  Poland | 10 | 9 | 15 | 7 | 41
  Brazil | 8 | 10 | 20 | 10 | 48
  Italy | 11 | 9 | 13 | 4 | 37
  France | 9 | 6 | 16 | 8 | 39
  Germany | 15 | 18 | 37 | 18 | 88
  Japan | 15 | 16 | 32 | 16 | 79
  Russia | 5 | 2 | 5 | 2 | 14
  Spain | 7 | 7 | 15 | 6 | 35
  Switzerland | 0 | 1 | 1 | 2 | 4
  United Kingdom | 4 | 5 | 6 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75) (Placebo, 2 mg or 4 mg Baricitinib)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All participants randomized to placebo, 2 mg or 4 mg of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 185 | 92
percentage of participants | 17.2 [10.9 to 26.1] | 27.6 [21.6 to 34.4] | 31.5 [22.9 to 41.6]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.071, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.95 to 3.32]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.07 to 4.30]

2. Secondary Outcome: Percentage of Participants Achieving EASI75 (Placebo, 1 mg Baricitinib)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
  Missing values were imputed using Non-Responder Imputation (NRI), where non-responders were participants who permanently discontinue, are rescued, or are without at least 1 post-baseline observation.
Time Frame: Week 16
Population: All participants randomized to placebo or 1 mg of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib
Number analyzed (Participants) | 93 | 93
percentage of participants | 17.2 [10.9 to 26.1] | 22.6 [15.3 to 32.1]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.427, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.65 to 2.77]

3. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1 With a ≥ 2 Point Improvement
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 9.7 [5.2 to 17.4] | 12.9 [7.5 to 21.2] | 15.1 [10.7 to 21.0] | 21.7 [14.5 to 31.2]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.513, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.55 to 3.35]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.242, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.73 to 3.53]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.030, Regression, Logistic; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.09 to 5.90]

4. Secondary Outcome: Percentage of Participants Achieving EASI90
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease). The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 6.5 [3.0 to 13.4] | 8.6 [4.4 to 16.1] | 10.3 [6.7 to 15.5] | 14.1 [8.4 to 22.7]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.611, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.45 to 3.83]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.325, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.63 to 3.99]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.100, Regression, Logistic; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.85 to 6.14]

5. Secondary Outcome: Percent Change From Baseline in EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease).
  Least Squares Mean (LSM) were calculated using mixed model repeated measures (MMRM) model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline score and baseline score-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EASI data.
Measure: Geometric Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 54 | 61 | 144 | 65
percent change | -42.69 (4.135) | -60.34 (4.018) | -56.05 (2.755) | -63.31 (3.922)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -17.65, 95% CI 2-sided [-28.71 to -6.58], Standard Error of Mean 5.627
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -13.35, 95% CI 2-sided [-22.83 to -3.87], Standard Error of Mean 4.820
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -20.62, 95% CI 2-sided [-31.54 to -9.70], Standard Error of Mean 5.554

6. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD75)
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with a visual analogue scales (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 1.1 [0.2 to 5.8] | 6.5 [3.0 to 13.4] | 8.1 [5.0 to 12.9] | 6.5 [3.0 to 13.5]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.115, Regression, Logistic; Odds Ratio (OR) = 4.14, 95% CI 2-sided [0.71 to 24.29]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 5.85, 95% CI 2-sided [1.11 to 30.88]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.083, Regression, Logistic; Odds Ratio (OR) = 4.78, 95% CI 2-sided [0.81 to 28.08]

7. Secondary Outcome: Percentage of Participants Achieving a 4-Point Improvement in Itch Numeric Rating Scale (NRS)
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: Week 16
Population: All randomized participants with a baseline Itch NRS score >=4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 85 | 78 | 166 | 76
percentage of participants | 8.2 [4.0 to 16.0] | 23.1 [15.1 to 33.6] | 22.9 [17.2 to 29.9] | 38.2 [28.1 to 49.4]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.29 to 8.32]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.71, 95% CI 2-sided [1.59 to 8.66]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.00002, Regression, Logistic; Odds Ratio (OR) = 6.85, 95% CI 2-sided [2.79 to 16.82]

8. Secondary Outcome: Change From Baseline in the Score of Item 2 of the Atopic Dermatitis Sleep Scale (ADSS)
Description: The ADSS is a 3-item, participant-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep due to itch, frequency of waking due to itch, and difficulty getting back to sleep last night due to itch. Item 2 frequency of waking last night is reported by selecting the number of times they woke up each night, ranging from 0 to 29 times, where the higher a number indicates a worse outcome. The ADSS is designed to be completed daily, using a daily diary, with respondents thinking about sleep "last night." Each item is scored individually.
  LS Mean were calculated using an MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 ADSS Item 2 (frequency of waking) data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 53 | 62 | 135 | 66
units on a scale | -0.63 (0.149) | -1.05 (0.142) | -0.85 (0.099) | -1.42 (0.140)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.039, Mixed Models Analysis; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.82 to -0.02], Standard Error of Mean 0.203
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.23, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.56 to 0.13], Standard Error of Mean 0.175
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.18 to -0.39], Standard Error of Mean 0.201

9. Secondary Outcome: Change From Baseline in Skin Pain NRS
Description: Skin Pain NRS is a participant-administered,11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number, using a daily diary, that best describes the worst level of skin pain in the past 24 hours.
  LS Mean were calculated using MMRM model includes treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 Skin Pain NRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 53 | 62 | 135 | 66
units on a scale | -1.56 (0.284) | -2.27 (0.274) | -2.40 (0.193) | -3.02 (0.271)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.0714, Mixed Models Analysis; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.47 to 0.06], Standard Error of Mean 0.388
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.0134, Mixed Models Analysis; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.50 to -0.17], Standard Error of Mean 0.337
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-2.21 to -0.69], Standard Error of Mean 0.386

10. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1 With a >=2-point Improvement
Description: as for outcome 3
Time Frame: Week 24
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 12.9 [7.5 to 21.2] | 20.4 [13.5 to 29.7] | 18.9 [13.9 to 25.2] | 13.0 [7.6 to 21.4]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.183, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.78 to 3.75]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.235, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.76 to 3.11]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.991, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.43 to 2.36]

11. Secondary Outcome: Percentage of Participants Achieving EASI50
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease). The EASI50 is defined as a ≥ 50% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 35.5 [26.5 to 45.6] | 45.2 [35.4 to 55.3] | 51.4 [44.2 to 58.5] | 52.2 [42.1 to 62.1]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.263, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.77 to 2.57]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.016, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.13 to 3.19]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.06 to 3.52]

12. Secondary Outcome: Percentage of Participants Achieving EASI75
Description: as for outcome 1
Time Frame: Week 24
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 17.2 [10.9 to 26.1] | 30.1 [21.7 to 40.1] | 27.6 [21.6 to 34.4] | 25.0 [17.3 to 34.7]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.058, Regression, Logistic; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.98 to 3.96]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.072, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.95 to 3.32]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.224, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.76 to 3.18]

13. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: as for outcome 3
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 0.00 [0.0 to 4.0] | 2.2 [0.6 to 7.5] | 1.1 [0.3 to 3.9] | 3.3 [1.1 to 9.2]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.265, Regression, Logistic; Odds Ratio (OR) = 5.03, 95% CI 2-sided [0.29 to 86.08]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.520, Regression, Logistic; Odds Ratio (OR) = 2.54, 95% CI 2-sided [0.15 to 43.09]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.164, Regression, Logistic; Odds Ratio (OR) = 7.17, 95% CI 2-sided [0.45 to 99.99]

14. Secondary Outcome: Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Mean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 SCORAD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 54 | 60 | 142 | 64
units on a scale | -21.98 (2.171) | -28.06 (2.097) | -28.54 (1.438) | -31.74 (2.052)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.040, Mixed Models Analysis; Mean Difference (Final Values) = -6.08, 95% CI 2-sided [-11.88 to -0.29], Standard Error of Mean 2.948
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -6.56, 95% CI 2-sided [-11.54 to -1.58], Standard Error of Mean 2.533
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -9.77, 95% CI 2-sided [-15.51 to -4.03], Standard Error of Mean 2.919

15. Secondary Outcome: Percentage of Participants Achieving SCORAD90
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with a visual analogue scales (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD90 responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
percentage of participants | 0.00 [0.0 to 4.0] | 2.2 [0.6 to 7.5] | 1.1 [0.3 to 3.9] | 2.2 [0.6 to 7.6]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.265, Regression, Logistic; Odds Ratio (OR) = 4.75, 95% CI 2-sided [0.31 to 73.93]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.511, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [0.16 to 38.40]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.253, Regression, Logistic; Odds Ratio (OR) = 4.95, 95% CI 2-sided [0.32 to 77.11]

16. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected
Description: The BSA affected by AD will be assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. The overall total percentage will be reported based off of all 4 body regions combined, after applying specific multipliers to the different body regions to account for the percent of the total BSA represented by each of the 4 regions. Use the percentage of skin affected for each region (0 to 100%) in EASI as follows: BSA Total = 0.1*BSAhead and neck + 0.3*BSAtrunk + 0.2* BSAupper limbs + 0.4*BSAlower limbs.
  LS Mean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 BSA data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 54 | 61 | 144 | 65
units on a scale | -19.76 (2.257) | -25.98 (2.178) | -25.26 (1.488) | -28.17 (2.125)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.044, Mixed Models Analysis; Mean Difference (Final Values) = -6.21, 95% CI 2-sided [-12.26 to -0.16], Standard Error of Mean 3.078
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.037, Mixed Models Analysis; Mean Difference (Final Values) = -5.50, 95% CI 2-sided [-10.67 to -0.32], Standard Error of Mean 2.632
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -8.41, 95% CI 2-sided [-14.37 to -2.45], Standard Error of Mean 3.030

17. Secondary Outcome: Percentage of Participants Developing Skin Infections Requiring Antibiotic Treatment
Description: Percentage of participants developing skin infections requiring antibiotic treatment.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug and who did not discontinue from the study for the reason of "Lost to Follow-up" at the first post-baseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 184 | 92
percentage of participants | 5.4 | 6.5 | 6.5 | 5.4
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p > .999, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.797, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p > .999, Fisher Exact

18. Secondary Outcome: Mean Number of Days Without Topical Corticosteroids (TCS) Use
Description: The ANCOVA model includes treatment, region, and baseline disease severity (IGA) as factors.
Time Frame: Week 16
Population: All randomized participants without use of TCS.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 92 | 178 | 89
days | 12.18 (3.39) | 20.80 (3.37) | 17.65 (2.53) | 19.43 (3.41)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.056, ANCOVA; Mean Difference (Final Values) = 8.62, 95% CI 2-sided [-0.22 to 17.45], Standard Error of Mean 4.49
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.164, ANCOVA; Mean Difference (Final Values) = 5.48, 95% CI 2-sided [-2.24 to 13.19], Standard Error of Mean 3.92
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.110, ANCOVA; Mean Difference (Final Values) = 7.25, 95% CI 2-sided [-1.66 to 16.15], Standard Error of Mean 4.53

19. Secondary Outcome: Mean Gram Quantity of Low and Moderate Potency Background Topical Corticosteroid (TCS) Used (Tube Weights)
Description: Average weights of full tubes were used to determine the dispensed weights for each region. Returned tubes were weighed with cap without carton to determine the amount of TCS in grams (g) used at each visit. Analysis was done via analysis of variance (ANOVA), with geographic region, baseline disease severity, and treatment as factors in the model.
Time Frame: Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
grams | 242.59 (27.60) | 194.53 (27.42) | 185.70 (20.67) | 171.17 (27.16)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.178, ANOVA; Mean Difference (Final Values) = -48.06, 95% CI 2-sided [-118.00 to 21.88], Standard Error of Mean 35.63
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.066, ANOVA; Mean Difference (Final Values) = -56.90, 95% CI 2-sided [-117.56 to 3.77], Standard Error of Mean 30.90
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.045, ANOVA; Mean Difference (Final Values) = -71.42, 95% CI 2-sided [-141.24 to -1.60], Standard Error of Mean 35.57

20. Secondary Outcome: Percent Change From Baseline in Itch NRS
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity, visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 Itch NRS data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: Placebo administered orally every day in combination with topical corticosteroids. Additional placebo administered orally to maintain the blind.
- 1 mg Baricitinib: 1 mg Baricitinib administered orally every day in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  .
- 2 mg Baricitinib: 2 mg Baricitinib administered orally every day in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
- 4 mg Baricitinib: 4 mg Baricitinib administered orally every day in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 53 | 62 | 135 | 66
percent change | -17.48 (4.835) | -28.80 (4.663) | -32.89 (3.258) | -37.24 (4.609)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.088, Mixed Models Analysis; Mean Difference (Final Values) = -11.32, 95% CI 2-sided [-24.33 to 1.70], Standard Error of Mean 6.620
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = -15.41, 95% CI 2-sided [-26.67 to -4.16], Standard Error of Mean 5.725
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -19.76, 95% CI 2-sided [-32.71 to -6.82], Standard Error of Mean 6.583

21. Secondary Outcome: Percent Change From Baseline in Itch NRS at Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: All randomized participants with Week 24 itch NRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 1 mg Baricitinib: 1 mg Baricitinib administered orally every day in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 35 | 50 | 108 | 54
units on a scale | -15.35 (5.349) | -29.35 (5.039) | -30.11 (3.495) | -33.16 (4.972)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.055, Mixed Models Analysis; Mean Difference (Final Values) = -14.00, 95% CI 2-sided [-28.28 to 0.28], Standard Error of Mean 7.263
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.020, Mixed Models Analysis; Mean Difference (Final Values) = -14.76, 95% CI 2-sided [-27.15 to -2.38], Standard Error of Mean 6.297
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = -17.82, 95% CI 2-sided [-32.01 to -3.62], Standard Error of Mean 7.216

22. Secondary Outcome: Change From Baseline in the Total Score of the Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
  LS Mean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by visit-interactions as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 POEM data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 1 mg Baricitinib: 1 mg Baricitinib administered once daily day in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
  .
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 55 | 62 | 145 | 67
units on a scale | -4.18 (0.907) | -6.24 (0.872) | -7.27 (0.602) | -9.27 (0.855)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.095, Mixed Models Analysis; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-4.47 to -0.36], Standard Error of Mean 1.229
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-5.16 to -1.01], Standard Error of Mean 1.057
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -5.09, 95% CI 2-sided [-7.48 to -2.70], Standard Error of Mean 1.216

23. Secondary Outcome: Change From Baseline in the Patient Global Impression of Severity - Atopic Dermatitis (PGI-S-AD) Score
Description: The PGI-S-AD is a single-item question asking the participant how they would rate their overall AD symptoms over the past 24 hours, using a daily diary. The 5 categories of responses are "(0) no symptoms", "(1) very mild", "(2) mild" "(3) moderate", and "(4) severe."
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 PGI-S-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 53 | 62 | 135 | 66
units on a scale | -0.49 (0.107) | -0.74 (0.103) | -0.77 (0.072) | -1.07 (0.101)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.53 to 0.04], Standard Error of Mean 0.146
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.52 to -0.02], Standard Error of Mean 0.126
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.86 to -0.29], Standard Error of Mean 0.145

24. Secondary Outcome: Change From Baseline on the Hospital Anxiety Depression Scale (HADS)
Description: The HADS is a participant-rated instrument used to assess both anxiety and depression. This instrument consists of 14 item questionnaire, each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
  LS Mean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 HADS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 55 | 62 | 145 | 67
units on a scale
  Anxiety | -0.48 (0.382) | -1.04 (0.366) | -1.59 (0.256) | -1.32 (0.362)
  Depression | -0.40 (0.383) | -0.69 (0.367) | -1.03 (0.256) | -1.57 (0.362)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Anxiety; Test type: Superiority; p = 0.272, Mixed Models Analysis; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.58 to 0.45], Standard Error of Mean 0.516
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Anxiety; Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-1.99 to -0.24], Standard Error of Mean 0.446
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Anxiety; Test type: Superiority; p = 0.099, Mixed Models Analysis; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.85 to 0.16], Standard Error of Mean 0.511
Statistical Analysis 4: Comparison: Placebo vs 1 mg Baricitinib; Depression; Test type: Superiority; p = 0.584, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.30 to 0.74], Standard Error of Mean 0.519
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; Depression; Test type: Superiority; p = 0.162, Mixed Models Analysis; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.51 to 0.25], Standard Error of Mean 0.448
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; Depression; Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.18 to -0.15], Standard Error of Mean 0.515

25. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI)
Description: The DLQI is a simple, participant-administered,10 question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the last "week." Response categories include "not at all," "a little," "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively, and unanswered or "not relevant" responses scored as "0." Scores range from 0 to 30 ("no impact on participant's life" to "extremely large effect on participant's life"), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 DLQI data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 55 | 62 | 145 | 67
units on a scale | -4.95 (0.752) | -6.18 (0.719) | -6.57 (0.494) | -7.95 (0.705)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.228, Mixed Models Analysis; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-3.23 to 0.77], Standard Error of Mean 1.018
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.065, Mixed Models Analysis; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-3.35 to 0.10], Standard Error of Mean 0.876
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-4.99 to -1.02], Standard Error of Mean 1.007

26. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment - Atopic Dermatitis (WPAI-AD) Questionnaire
Description: The WPAI-AD participant questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. The WPAI-AD consists of 6 items grouped in 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment, that range from 0% to 100%, with higher values indicating greater impairment.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 WPAI-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 55 | 62 | 145 | 67
units on a scale
  Absenteeism: number analyzed (Participants) | 37 | 36 | 85 | 42
  Absenteeism | -4.77 (2.365) | -5.69 (2.433) | -2.98 (1.639) | -4.56 (2.258)
  Presenteeism: number analyzed (Participants) | 34 | 35 | 83 | 39
  Presenteeism | -14.86 (3.182) | -11.80 (3.161) | -14.56 (2.133) | -14.81 (3.000)
  Work Productivity Loss: number analyzed (Participants) | 34 | 35 | 83 | 39
  Work Productivity Loss | -13.22 (3.560) | -12.07 (3.565) | -13.07 (2.440) | -14.12 (3.396)
  Activity Impairment | -16.46 (2.853) | -18.46 (2.729) | -20.86 (1.847) | -23.92 (2.660)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Change from Baseline (CFB) Absenteeism; Test type: Superiority; p = 0.784, Mixed Models Analysis; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-7.50 to 5.67], Standard Error of Mean 3.339
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; CFB Absenteeism; Test type: Superiority; p = 0.525, Mixed Models Analysis; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [-3.75 to 7.34], Standard Error of Mean 2.813
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; CFB Absenteeism; Test type: Superiority; p = 0.947, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-6.11 to 6.53], Standard Error of Mean 3.204
Statistical Analysis 4: Comparison: Placebo vs 1 mg Baricitinib; CFB Presenteeism; Test type: Superiority; p = 0.488, Mixed Models Analysis; Mean Difference (Final Values) = 3.06, 95% CI 2-sided [-5.62 to 11.74], Standard Error of Mean 4.409
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; CFB Presenteeism; Test type: Superiority; p = 0.936, Mixed Models Analysis; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-7.02 to 7.62], Standard Error of Mean 3.720
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; CFB Presenteeism; Test type: Superiority; p = 0.991, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-8.35 to 8.45], Standard Error of Mean 4.267
Statistical Analysis 7: Comparison: Placebo vs 1 mg Baricitinib; CFB Work Productivity Loss; Test type: Superiority; p = 0.816, Mixed Models Analysis; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-8.57 to 10.88], Standard Error of Mean 4.938
Statistical Analysis 8: Comparison: Placebo vs 2 mg Baricitinib; CFB Work Productivity Loss; Test type: Superiority; p = 0.971, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-8.08 to 8.38], Standard Error of Mean 4.178
Statistical Analysis 9: Comparison: Placebo vs 4 mg Baricitinib; CFB Work Productivity Loss; Test type: Superiority; p = 0.852, Mixed Models Analysis; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-10.36 to 8.56], Standard Error of Mean 4.804
Statistical Analysis 10: Comparison: Placebo vs 1 mg Baricitinib; CFB Activity Impairment; Test type: Superiority; p = 0.607, Mixed Models Analysis; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-9.61 to 5.63], Standard Error of Mean 3.877
Statistical Analysis 11: Comparison: Placebo vs 2 mg Baricitinib; CFB Activity Impairment; Test type: Superiority; p = 0.186, Mixed Models Analysis; Mean Difference (Final Values) = -4.40, 95% CI 2-sided [-10.92 to 2.12], Standard Error of Mean 3.319
Statistical Analysis 12: Comparison: Placebo vs 4 mg Baricitinib; CFB Activity Impairment; Test type: Superiority; p = 0.052, Mixed Models Analysis; Mean Difference (Final Values) = -7.45, 95% CI 2-sided [-14.96 to 0.06], Standard Error of Mean 3.820

27. Secondary Outcome: Change From Baseline in the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Index Score United States and United Kingdom Algorithm
Description: The EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1, with higher score indicating better health state.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with EQ-5D-5L US and UK Health scores.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 55 | 62 | 145 | 67
units on a scale
  US Health State Index | 0.04 (0.016) | 0.08 (0.016) | 0.09 (0.011) | 0.11 (0.015)
  UK Health State Index | 0.06 (0.023) | 0.11 (0.022) | 0.13 (0.016) | 0.15 (0.022)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; CFB US Health State Index; Test type: Superiority; p = 0.131, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.08], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; CFB US Health State Index; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.01 to 0.08], Standard Error of Mean 0.019
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; CFB US Health State Index; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [0.02 to 0.11], Standard Error of Mean 0.022
Statistical Analysis 4: Comparison: Placebo vs 1 mg Baricitinib; CFB UK Health State Index; Test type: Superiority; p = 0.102, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.01 to 0.11], Standard Error of Mean 0.031
Statistical Analysis 5: Comparison: Placebo vs 2 mg Baricitinib; CFB UK Health State Index; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.01 to 0.12], Standard Error of Mean 0.027
Statistical Analysis 6: Comparison: Placebo vs 4 mg Baricitinib; CFB UK Health State Index; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.03 to 0.15], Standard Error of Mean 0.031

28. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Visual Analog Score (VAS)
Description: EQ-5D-5L is a 2-part measurement. The second part is assessed using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
  LS Means were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interactions as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EQ-5D-5L VAS data.
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 55 | 62 | 145 | 67
millimeters (mm) | 7.64 (2.407) | 11.63 (2.306) | 8.76 (1.588) | 11.03 (2.260)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.221, Mixed Models Analysis; Mean Difference (Final Values) = 3.99, 95% CI 2-sided [-2.41 to 10.39], Standard Error of Mean 3.256
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.689, Mixed Models Analysis; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-4.40 to 6.65], Standard Error of Mean 2.807
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.294, Mixed Models Analysis; Mean Difference (Final Values) = 3.39, 95% CI 2-sided [-2.95 to 9.74], Standard Error of Mean 3.226

29. Secondary Outcome: Percentage of Participants Achieving EASI75
Description: as for outcome 1
Time Frame: Week 52
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 1 mg Baricitinib: 1 mg Baricitinib administered once daily day in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 93 | 93 | 185 | 92
Percentage of participants | 26.9 [18.9 to 36.7] | 33.3 [24.6 to 43.4] | 30.3 [24.1 to 37.2] | 37.0 [27.8 to 47.2]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.382, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.70 to 2.54]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.638, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.65 to 2.02]
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.169, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.83 to 2.96]

30. Secondary Outcome: Percent Change From Baseline in Itch NRS at Week 52
Description: as for outcome 20
Time Frame: Baseline, Week 52
Population: All randomized participants with Week 52 Itch NRS data.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 44 | 54 | 110 | 56
Percent Change | -12.13 (7.075) | -19.49 (6.679) | -16.01 (4.729) | -29.31 (6.619)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.447, Regression, Linear; LS Mean Difference (Final Values) = -7.36, 95% CI 2-sided [-26.38 to 11.66], Standard Error of Mean 9.674
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.646, Regression, Linear; LS Mean Difference (Final Values) = -3.88, 95% CI 2-sided [-20.50 to 12.74], Standard Error of Mean 8.454
Statistical Analysis 3: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.075, Regression, Linear; LS Mean Difference (Final Values) = -17.18, 95% CI 2-sided [-36.14 to 1.77], Standard Error of Mean 9.640

31. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at 16 Weeks After Rerandomization (Week 68) Randomized Downtitration (All Participants Entering the Substudy)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. All missing values were imputed using modified last observation carried forward (mLOCF).
Time Frame: Week 68
Population: Participants who received at least one study medication during Week 52 to Week 200 in Study JAIN and entered the downtitration substudy. Additionally, those participants who did not meet study discontinuation criteria and continued will be considered in the analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders): 4 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 16 | 16 | 25 | 24
Percentage of participants | 93.8 [71.7 to 98.9] | 56.3 [33.2 to 76.9] | 84.0 [65.3 to 93.6] | 50.0 [31.4 to 68.6]

32. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at 16 Weeks After Rerandomization (Week 104) Randomized Downtitration (All Participants Entering the Substudy)
Description: as for outcome 31
Time Frame: Week 104
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 16 | 16 | 25 | 24
Percentage of participants | 68.8 [44.4 to 85.8] | 50.0 [28.0 to 72.0] | 72.0 [52.4 to 85.7] | 25.0 [12.0 to 44.9]

33. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1 Assessed at 16 Weeks After Rerandomization (Week 68) Randomized Downtitration (All Participants Entering the Substudy)
Description: as for outcome 3
Time Frame: Week 68
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- LTE Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders): 4 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | LTE Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 16 | 16 | 25 | 24
Percentage of participants | 50 [28.0 to 72.0] | 25.0 [10.2 to 49.5] | 44.0 [26.7 to 62.9] | 20.8 [9.2 to 40.5]

34. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1 Assessed at 16 Weeks After Rerandomization (Week 104) Randomized Downtitration (All Participants Entering the Substudy)
Description: as for outcome 3
Time Frame: Week 104
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 16 | 16 | 25 | 24
Percentage of participants | 43.8 [23.1 to 66.8] | 25.0 [10.2 to 49.5] | 44.0 [26.7 to 62.9] | 8.3 [2.3 to 25.8]

35. Secondary Outcome: Percentage of Participants With a Response of EASI75 From Baseline Assessed at 16 Weeks After Rerandomization (Week 68) Randomized Downtitration (All Participants Entering the Substudy)
Description: as for outcome 1
Time Frame: Week 68
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 16 | 16 | 25 | 24
Percentage of participants | 75.0 [50.5 to 89.8] | 56.3 [33.2 to 76.90] | 72.0 [52.4 to 85.7] | 41.7 [24.5 to 61.2]

36. Secondary Outcome: Percentage of Participants With a Response of EASI75 From Baseline Assessed at 16 Weeks After Rerandomization (Week 104) Randomized Downtitration (All Participants Entering the Substudy)
Description: as for outcome 1
Time Frame: Week 104
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4mg Baricitinib to 4mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 16 | 16 | 25 | 24
Percentage of participants | 68.8 [44.4 to 85.8] | 56.3 [33.2 to 76.9] | 56.0 [37.1 to 73.3] | 33.3 [18.0 to 53.3]

37. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at 16 Weeks After Rerandomization (Week 68) Randomized Downtitration (Participants Entering the Substudy With IGA 0 or 1)
Description: as for outcome 31
Time Frame: Week 68
Population: Participants who received at least one study medication during Week 52 to Week 200 in Study JAIN and entered the downtitration substudy with IGA 0 or 1 at Week 52. Additionally, those participants who did not meet study discontinuation criteria and continued will be considered in the analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- LTE Substudy 4mg Baricitinib to 4mg Baricitinib(Responders/Partial Responders): 4 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | LTE Substudy 4mg Baricitinib to 4mg Baricitinib(Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 10 | 9 | 10 | 9
Percentage of participants | 100 [72.2 to 100] | 77.8 [45.3 to 93.7] | 100 [72.2 to 100] | 55.6 [26.7 to 81.1]

38. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at 16 Weeks After Rerandomization (Week 104) Randomized Downtitration (Participants Entering the Substudy With IGA 0 or 1)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. All missing values were imputed using mLOCF.
Time Frame: Week 104
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 10 | 9 | 10 | 9
Percentage of participants | 80.0 [49.0 to 94.3] | 66.7 [35.4 to 87.9] | 100 [72.2 to 100] | 33.3 [12.1 to 64.6]

39. Secondary Outcome: Percentage of Participants With a Response of IGA 0 or 1 Assessed at 16 Weeks After Rerandomization (Week 68) Randomized Downtitration (Participants Entering the Substudy With IGA 0 or 1)
Description: as for outcome 38
Time Frame: Week 68
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 10 | 9 | 10 | 9
Percentage of participants | 60.0 [31.3 to 83.2] | 33.3 [12.1 to 64.6] | 90.0 [59.6 to 98.2] | 55.6 [26.7 to 81.1]

40. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1 Assessed at 16 Weeks After Rerandomization (Week 104) Randomized Downtitration (Participants Entering the Substudy With IGA 0 or 1)
Description: as for outcome 38
Time Frame: Week 104
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 1 mg Baricitinib (Responders/Partial Responders)
Number analyzed (Participants) | 10 | 9 | 10 | 9
Percentage of participants | 50.0 [23.7 to 76.3] | 33.3 [12.1 to 64.6] | 90.0 [59.6 to 98.2] | 22.2 [6.3 to 54.7]

41. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at Week 68 Participants Not Entered Into Substudy (All Participants)
Description: as for outcome 38
Time Frame: Week 68
Population: Participants who received at least one study medication Week 52 to Week 200 in Study JAIN, and were Responders (IGA 0 or 1) and Partial Responders (IGA 2) at Week 52 but were not eligible for downtitration substudy (i.e. had study drug interrupted at Week 52, or had received high or ultra-high potency TCS in the previous 14 days). Additionally, those participants who did not met study discontinuation criteria and continued will be considered in the analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- LTE 1 mg Baricitinib (Responders/ Partial Responders) - Did Not Enter Substudy: 1 mg administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/ Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy
Number analyzed (Participants) | 7 | 22 | 34 | 29
Percentage of participants | 100 [64.6 to 100] | 86.4 [66.7 to 95.3] | 100 [89.8 to 100] | 93.1 [78.0 to 98.1]

42. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at Week 104 Participants Not Entered Into Substudy (All Participants)
Description: as for outcome 38
Time Frame: Week 104
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy
Number analyzed (Participants) | 7 | 22 | 34 | 29
Percentage of participants | 100 [64.6 to 100] | 86.4 [66.7 to 95.3] | 97.1 [85.1 to 99.5] | 93.1 [78.0 to 98.1]

43. Secondary Outcome: Percentage of Participants With a Response of IGA 0 or 1 Assessed at Week 68 - Participants Not Entered Into Substudy (All Participants)
Description: as for outcome 38
Time Frame: Week 68
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy
Number analyzed (Participants) | 7 | 22 | 34 | 29
Percentage of participants | 14.3 [2.6 to 51.3] | 50.0 [30.7 to 69.3] | 47.1 [31.5 to 63.3] | 51.7 [34.4 to 68.6]

44. Secondary Outcome: Percentage of Participants With a Response of IGA 0 or 1 Assessed at Week 104 - Participants Not Entered Into Substudy (All Participants)
Description: as for outcome 38
Time Frame: Week 104
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy
Number analyzed (Participants) | 7 | 22 | 34 | 29
Percentage of participants | 42.9 [15.8 to 75.0] | 50.0 [30.7 to 69.3] | 47.1 [31.5 to 63.3] | 48.3 [31.4 to 65.6]

45. Secondary Outcome: Percentage of Participants With A Response of EASI75 Assessed at Week 68 - Participants Not Entered Into Substudy (All Participants)
Description: as for outcome 1
Time Frame: Week 68
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy
Number analyzed (Participants) | 7 | 22 | 34 | 29
Percentage of participants | 57.1 [25.0 to 84.2] | 63.6 [43.0 to 80.3] | 76.5 [60.0 to 87.6] | 62.1 [44.0 to 77.3]

46. Secondary Outcome: Percentage of Participants With A Response of EASI75 Assessed at Week 104 - Participants Not Entered Into Substudy (All Participants)
Description: as for outcome 1
Time Frame: Week 104
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy
Number analyzed (Participants) | 7 | 22 | 34 | 29
Percentage of participants | 85.7 [48.7 to 97.4] | 68.2 [47.3 to 83.6] | 70.6 [53.8 to 83.2] | 72.4 [54.3 to 85.3]

47. Secondary Outcome: Time to Retreatment (Time to IGA ≥3) Randomized Downtitration (All Patients Entering the Substudy)
Description: Participants who entered the Substudy and relapsed with an IGA ≥3.
Time Frame: Week 52 Up to Week 200
Population: Participants who received at least one study medication during Week 52 to Week 200 in Study JAIN, entered the downtitration substudy and experienced relapse from Week 52 up to Week 200. Additionally, those participants who did not meet study discontinuation criteria and continued will be considered in the analysis set.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- 4 mg Baricitinib to 4 mg Baricitinib to 4 mg Baricitinib: 4 mg Baricitinib participants randomized to 4 mg Baricitinib in the downtitration substudy who experienced worsening symptoms (IGA increased to ≥3), were retreated with their presubstudy 4 mg Baricitinib dose.
- 4 mg Baricitinib to 2 mg Baricitinib to 4 mg Baricitinib: 4 mg Baricitinb participants randomized to 2 mg Baricitinib in the downtitration substudy who experienced worsening symptoms (IGA increased to ≥3), were retreated with their presubstudy 4 mg Baricitinib dose.
- 2 mg Baricitinib to 2 mg Baricitinib to 2 mg Baricitinib: 2 mg Baricitinb participants randomized to 2 mg Baricitinib in the downtitration substudy who experienced worsening symptoms (IGA increased to ≥3), were retreated with their presubstudy 2 mg Baricitinib dose.
- 2 mg Baricitinib to 1 mg Baricitinib to 2 mg Baricitinib: 2 mg Baricitinib participants randomized to 1 mg Baricitinib in the downtitration substudy who experienced worsening symptoms (IGA increased to ≥3), were retreated with their presubstudy 2 mg Baricitinib dose.
Arm/Group | 4 mg Baricitinib to 4 mg Baricitinib to 4 mg Baricitinib | 4 mg Baricitinib to 2 mg Baricitinib to 4 mg Baricitinib | 2 mg Baricitinib to 2 mg Baricitinib to 2 mg Baricitinib | 2 mg Baricitinib to 1 mg Baricitinib to 2 mg Baricitinib
Number analyzed (Participants) | 5 | 11 | 15 | 20
Days | 218 [29 to NA] — Upper Confidence Level (CI) not estimable due to censoring. | 79 [28 to 359] | 68 [28 to 364] | 71 [29 to 225]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 200
Description: All randomized participants who received at least 1 dose of investigational product and who did not discontinue from the study for the reason 'Lost to Follow-up' at the first postbaseline visit. This definition excludes participants with no safety assessments postbaseline so that incidence rates are not underestimated. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Long Term Extension(LTE) Substudy 2mg Baricitinib to 1mg Baricitinib (Responders/Partial Responders): 2 mg Baricitinib rerandomized to 1 mg Baricitinib administered orally once daily in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
- LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy: Placebo rerandomized to 4 mg Baricitinib administered orally once daily (continued previous dose) in combination with topical corticosteroids. Placebo administered orally to maintain the blind.
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | 4 mg Baricitinib | Long Term Extension(LTE) Substudy 2mg Baricitinib to 1mg Baricitinib (Responders/Partial Responders) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy | LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy | LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93 | 0/185 | 0/92 | 0/24 | 0/25 | 0/16 | 0/16 | 0/29 | 0/34 | 0/22 | 0/7 | 0/11 | 0/12 | 0/13 | 0/14 | 0/27 | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 5/93 | 7/93 | 9/184 | 10/92 | 3/24 | 4/25 | 3/16 | 3/16 | 1/29 | 1/34 | 1/22 | 2/7 | 1/11 | 2/12 | 2/13 | 3/14 | 3/27 | 5/26 | 4/24
Other Adverse Events (participants affected / at risk) | 50/93 | 63/93 | 130/184 | 75/92 | 17/24 | 16/25 | 13/16 | 16/16 | 16/29 | 25/34 | 16/22 | 7/7 | 6/11 | 10/12 | 11/13 | 13/14 | 18/27 | 18/26 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=93) | 1 mg Baricitinib (N=93) | 2 mg Baricitinib (N=184) | 4 mg Baricitinib (N=92) | Long Term Extension(LTE) Substudy 2mg Baricitinib to 1mg Baricitinib (Responders/Partial Responders) (N=24) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) (N=25) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) (N=16) | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) (N=16) | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy (N=29) | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (N=34) | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (N=22) | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (N=7) | LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=11) | LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=12) | LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=13) | LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=14) | LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=27) | LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=26) | LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=24)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/49 (0) | 0/58 (0) | 0/132 (0) | 0/57 (0) | 0/21 (0) | 0/20 (0) | 0/10 (0) | 0/8 (0) | 0/15 (0) | 0/21 (0) | 0/14 (0) | 0/3 (0) | 0/4 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/20 (0) | 0/20 (0) | 0/17 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=93) | 1 mg Baricitinib (N=93) | 2 mg Baricitinib (N=184) | 4 mg Baricitinib (N=92) | Long Term Extension(LTE) Substudy 2mg Baricitinib to 1mg Baricitinib (Responders/Partial Responders) (N=24) | LTE Substudy 2 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) (N=25) | LTE Substudy 4 mg Baricitinib to 2 mg Baricitinib (Responders/Partial Responders) (N=16) | LTE Substudy 4 mg Baricitinib to 4 mg Baricitinib (Responders/Partial Responders) (N=16) | LTE Placebo (Responders/Partial Responders) - Did Not Enter Substudy (N=29) | LTE 1 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (N=34) | LTE 2 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (N=22) | LTE 4 mg Baricitinib (Responders/Partial Responders) - Did Not Enter Substudy (N=7) | LTE Placebo to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=11) | LTE Placebo to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=12) | LTE 1 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=13) | LTE 1 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=14) | LTE 2 mg Baricitinib to 2 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=27) | LTE 2 mg Baricitinib to 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=26) | LTE 4 mg Baricitinib (Non-responders) - Did Not Enter Substudy (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratoconus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (3) | 7 (7) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 9 (10) | 6 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (11) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 0 (0) | 6 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (3) | 1 (1) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (3) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 1 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 1 (1) | 4 (4) | 4 (5) | 6 (6) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 5 (5) | 4 (5)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ear infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 2 (4) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0) | 4 (5) | 4 (5) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 2 (3) | 9 (11) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (3) | 1 (3)
Furuncle (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (2) | 1 (1) | 5 (5) | 6 (7) | 2 (2) | 1 (2) | 0 (0) | 3 (5) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 4 (4) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (4) | 15 (18) | 14 (15) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 14 (25) | 16 (20) | 36 (48) | 34 (45) | 8 (11) | 3 (4) | 3 (3) | 3 (7) | 3 (3) | 4 (5) | 5 (5) | 4 (5) | 1 (2) | 6 (7) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 2 (3)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 6 (6) | 5 (7) | 6 (9) | 7 (13) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (3) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Perichondritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-acute covid-19 syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 6 (6) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 3 (4) | 4 (4) | 4 (5) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (5) | 7 (10) | 4 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (7) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1/44 (1) | 0/35 (0) | 0/52 (0) | 0/35 (0) | 0/3 (0) | 0/5 (0) | 0/6 (0) | 0/8 (0) | 1/14 (1) | 0/13 (0) | 0/8 (0) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0) | 0/7 (0) | 0/6 (0) | 0/7 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/44 (0) | 0/35 (0) | 2/52 (2) | 0/35 (0) | 0/3 (0) | 1/5 (1) | 0/6 (0) | 0/8 (0) | 0/14 (0) | 1/13 (1) | 1/8 (1) | 1/4 (1) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0) | 1/7 (1) | 0/6 (0) | 0/7 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (5)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthroscopy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0/49 (0) | 0/58 (0) | 0/132 (0) | 0/57 (0) | 0/21 (0) | 0/20 (0) | 0/10 (0) | 0/8 (0) | 0/15 (0) | 0/21 (0) | 0/14 (0) | 0/3 (0) | 0/4 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/20 (0) | 0/20 (0) | 0/17 (0)
Sars-cov-2 antibody test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 7 (8) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (9) | 6 (7) | 6 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 8 (15) | 14 (17) | 10 (13) | 1 (2) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (3) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Premature ejaculation (Psychiatric disorders) | 0/49 (0) | 0/58 (0) | 0/132 (0) | 0/57 (0) | 0/21 (0) | 0/20 (0) | 0/10 (0) | 0/8 (0) | 0/15 (0) | 0/21 (0) | 1/14 (1) | 0/3 (0) | 0/4 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/20 (0) | 0/20 (0) | 0/17 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/44 (0) | 0/35 (0) | 0/52 (0) | 0/35 (0) | 0/3 (0) | 0/5 (0) | 0/6 (0) | 0/8 (0) | 0/14 (0) | 0/13 (0) | 1/8 (1) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0) | 0/7 (0) | 0/6 (0) | 0/7 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/44 (0) | 2/35 (3) | 0/52 (0) | 0/35 (0) | 0/3 (0) | 0/5 (0) | 0/6 (0) | 0/8 (0) | 0/14 (0) | 3/13 (9) | 0/8 (0) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0) | 0/7 (0) | 0/6 (0) | 1/7 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/44 (0) | 0/35 (0) | 0/52 (0) | 0/35 (0) | 0/3 (0) | 0/5 (0) | 0/6 (0) | 0/8 (0) | 0/14 (0) | 1/13 (1) | 0/8 (0) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0) | 0/7 (0) | 0/6 (0) | 0/7 (0)
Prostatitis (Reproductive system and breast disorders) | 0/49 (0) | 0/58 (0) | 0/132 (0) | 0/57 (0) | 1/21 (1) | 0/20 (0) | 0/10 (0) | 0/8 (0) | 0/15 (0) | 0/21 (0) | 0/14 (0) | 0/3 (0) | 0/4 (0) | 0/9 (0) | 1/9 (1) | 0/8 (0) | 0/20 (0) | 0/20 (0) | 0/17 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0/44 (0) | 0/35 (0) | 0/52 (0) | 0/35 (0) | 0/3 (0) | 0/5 (0) | 0/6 (0) | 1/8 (1) | 0/14 (0) | 0/13 (0) | 0/8 (0) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0) | 0/7 (0) | 0/6 (0) | 0/7 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 3 (4) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 9 (10) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (10) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intrauterine contraception (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0/49 (0) | 0/58 (0) | 0/132 (0) | 0/57 (0) | 0/21 (0) | 0/20 (0) | 0/10 (0) | 0/8 (0) | 0/15 (0) | 0/21 (0) | 0/14 (0) | 0/3 (0) | 0/4 (0) | 0/9 (0) | 0/9 (0) | 1/8 (1) | 0/20 (0) | 0/20 (0) | 0/17 (0)
Retinopexy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tooth restoration (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polypectomy (Surgical and medical procedures) | 0/44 (0) | 0/35 (0) | 0/52 (0) | 0/35 (0) | 0/3 (0) | 0/5 (0) | 0/6 (0) | 0/8 (0) | 0/14 (0) | 0/13 (0) | 0/8 (0) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/4 (0) | 1/6 (1) | 0/7 (0) | 0/6 (0) | 0/7 (0)
Vasectomy (Surgical and medical procedures) | 0/49 (0) | 0/58 (0) | 0/132 (0) | 0/57 (0) | 0/21 (0) | 0/20 (0) | 1/10 (1) | 0/8 (0) | 0/15 (0) | 0/21 (0) | 0/14 (0) | 0/3 (0) | 0/4 (0) | 0/9 (0) | 0/9 (0) | 0/8 (0) | 0/20 (0) | 0/20 (0) | 0/17 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 5 (5) | 3 (3) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03428100/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03428100/SAP_002.pdf